CLINICAL TRIAL: NCT03119662
Title: Parallel-Group, Placebo-Controlled Randomized Study Investigating the Effect of Intravenous Iso-osmolar Iodinated Contrast Material Iodixanol (Visipaque™ Injection 320 mgI/mL) on Renal Function in Adults With Chronic Kidney Disease (CKD) Stage III or Stage IV Who Have Undergone Endovascular Aneurysm Repair (EVAR)
Brief Title: A Study to Explore the Renal Safety of Visipaque Injection 320 mgI/mL in Patients With Chronic Kidney Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was discontinued due to a lower than anticipated recruitment rate. The decision has not been made due to any safety reasons.
Sponsor: GE Healthcare (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GE-012-106; 2016-001668-13 (EudraCT Number)
Record Dates: First submitted 2017-03-21; First posted 2017-04-18 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-11

CONDITIONS: Chronic Kidney Diseases
Keywords: Acute kidney injury (AKI); Acute kidney injury network (AKIN); Chronic kidney disease (CKD); Contrast-enhanced computed tomography (CECT); Endovascular Aneurysm Repair (EVAR); Iodixanol; Non-enhanced computed tomography (NECT); Serum creatinine (SCr)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury | interventions — iodixanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Visipaque™: Contrast-Enhanced Computed Tomography (CECT) (Experimental): Participants received 1 intravenous injection of Visipaque™ 320 mg I/ml injection (100 mL iodixanol) and underwent computed tomography (CT) examination.
  Interventions: Drug: Visipaque
- Saline: Non-Enhanced Computed Tomography (NECT) (Placebo Comparator): Participants received 1 intravenous injection of saline placebo (matched to Visipaque™ 320 mg I/ml injection) and underwent computed tomography (CT) examination and supplemental non-contrast duplex ultrasonography imaging examination.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Visipaque — 100 mL iodixanol (Visipaque Injection 320 mg I/mL), followed by a 10 mL saline flush to ensure delivery of the full dose of Visipaque.
  Arms: Visipaque™: Contrast-Enhanced Computed Tomography (CECT)
Drug: Placebos — 100 mL saline, followed by a 10 mL saline flush.
  Arms: Saline: Non-Enhanced Computed Tomography (NECT)

SUMMARY:
This parallel-group, randomized, placebo-controlled study will examine the incidence and severity of acute kidney injury (AKI) in patients with chronic kidney disease (CKD) stage III/IV following an i.v. injection of iso-osmolar iodinated contrast material iodixanol (Visipaque™ Injection 320 mgI/mL), as compared with patients who received saline and underwent a non-enhanced CT (NECT) and duplex ultrasound (US) during their scheduled post-EVAR surveillance imaging.

DETAILED DESCRIPTION:
GEHC has decided not to provide this detail

ELIGIBILITY:
Inclusion Criteria:

* Was ≥18 years of age at the time that written informed consent is obtained.
* Was male or is a nonpregnant, nonlactating female who is either surgically sterile or is postmenopausal. Women of childbearing potential must use adequate contraception from Screening until 30 days after the Baseline Visit and must have a negative pregnancy test at the Baseline Visit.
* Was an outpatient who has undergone successful EVAR and is scheduled for his/her next post-procedural imaging follow-up examination.
* Had previously completed one or more of his or her post-EVAR surveillance imaging examination(s) that provided evidence on stable post-EVAR status.
* Had a documented diagnosis of stage III or IV CKD and stable renal function.
* Was able to provide written informed consent.
* Was able and willing to comply with all study procedures as described in the protocol.

Exclusion Criteria:

* Was pregnant, lactating, is possibly pregnant, or is actively trying to conceive during the study period.
* Was a patient for whom an endoleak or other clinically meaningful EVAR-related complication (as judged by the investigator) has already been discovered.
* Was undergoing surveillance following a Thoracic Endovascular Repair (TEVAR).
* Had a known or suspected history of immediate or delayed hypersensitivity to iodine or any iodinated contrast medium.
* Was using metformin (e.g., Glucophage®) that cannot be discontinued for the period of 24 hours prior to the Baseline Visit and for at least 48 hours after the imaging procedure.
* Had been exposed to any intravascular iodinated contrast medium in the 7 days prior to the Baseline Visit.
* Had congestive heart failure (New York Heart Association [NYHA] Class IV) or hepatic failure/liver cirrhosis.
* Had Stage V CKD.
* Had a pre-existing requirement for renal dialysis.
* Had undergone percutaneous transluminal renal angioplasty (PTRA) within 12 months before the index EVAR procedure or is scheduled to undergo PTRA during the study period.
* Had any clinically active, serious, life-threatening disease, medical, or significant psychiatric condition; has a life expectancy of less than 6 months; or is, in the Investigator's opinion, unsuitable for participation in the study for any reason.
* Had been enrolled in another clinical study within the 30 days prior to the Screening Visit or is planned to enroll in another clinical study within the duration of this study.
* Had been previously enrolled in this study.
* Was using i.v. vasopressor or inotropic medications.
* Had used nonsteroidal anti-inflammatory drugs (NSAIDs) or any nephrotoxic medication within 48 hours of the Baseline Visit or will do so within 72 hours after the CT procedure-with the exception of acetylsalicylic acid (Aspirin) at a dose of ≤100 mg daily (QD).
* Had been hospitalized within 30 days prior to Screening Visit for any reason other than practical purposes for management of tests or diagnostic assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (17):
  - University Hospital, Birmingham, Alabama
  - : Aventiv Research Inc., Mesa, Arizona
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Alliance Research Centers, Laguna Hills, California
  - Universal Axon Clinical Research, LLC, Doral, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University of South Florida - South Tampa Campus, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Hospital, Louisville, Kentucky
  - Boston University Medical Center/Boston Medical Center, Boston, Massachusetts
  - The Duluth Clinic, Ltd., Duluth, Minnesota
  - Mount Sinai West, New York, New York
  - University of North Carolina at Chapel Hill Clinical Translational Research Center, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - CRCHUM- CHUM Research Center, Montreal
  - St. Boniface General Hospital, Winnipeg
- Poland (4):
  - Oddzial Chirurgii Naczyniowej i Ogolnej, Wojewodzki Szpital Specjalistyczny Nr 4 w Bytomiu, Bytom
  - Klinika Kardiochirurgii i Chirurgii Naczyniowej, Uniwersyteckie Centrum Kliniczne, Gdansk
  - Klinika Chirurgii Naczyniowej i Angiologii, Samodzielny Publiczny Szpital Kliniczny nr 1, Lublin
  - Oddzial Chirurgii Ogolnej i Naczyn, Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego, Poznan
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Son Espases, Palma
- United Kingdom (2):
  - St. George's Healthcare NHS Trust, St. George's Hospital, London
  - Royal Stoke University Hospital, Radiology Department, Stoke-on-Trent

REFERENCES:
- [Derived] Solomon R. PRESERVE: The End or the Beginning of a New Era in Prevention of Contrast-Associated Acute Kidney Injury? Am J Kidney Dis. 2018 Sep;72(3):322-324. doi: 10.1053/j.ajkd.2018.03.013. Epub 2018 May 8. No abstract available. PMID 29751980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Study was conducted at 29 sites in United States of America & Europe from 8 February 2018 to 19 October 2018. A total of 4 participants with Chronic Kidney Disease (CKD) stage III/IV were enrolled in the study.
Pre-assignment Details: Participants were randomized in 1:1 ratio to undergo either contrast-enhanced computed tomography (CECT) or non-enhanced computed tomography (NECT), of which 1 participant withdrew from study.
Period: Overall Study
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Visipaque™: Contrast-Enhanced Computed Tomography (CECT): Participants received 1 intravenous injection of Visipaque™ 320 mg I/ml injection (100 mL iodixanol) and underwent CT examination.
- Saline: Non-Enhanced Computed Tomography (NECT): Participants received 1 intravenous injection of saline placebo (matched to Visipaque™ 320 mg I/ml injection) and underwent CT examination and supplemental non-contrast duplex ultrasonography imaging examination.
- Total: Total of all reporting groups
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Incidence of Acute Kidney Injury (AKI) Stage >=1 Per Acute Kidney Injury Network (AKIN) Serum Creatinine (SCr) Criteria
Description: AKIN Serum Creatinine Criteria for AKI- Stage 1: a SCr increase of >=0.3 mg/dL (>=26.4 μmol/L) or increase to >=150% to 200% (>=1.5- to 2.0-fold) from baseline within 48 hours. Stage 2: a SCr increase to >200% to 300% (>2.0- to 3-fold) from baseline within 48 hours. Stage 3: a SCr increase to >300% (>3.0-fold) from baseline or SCr >=4.0 mg/dL (>=354 μmol/L) with an acute increase of >=0.5 mg/dL (>=44 μmol/L) within 48 hours.
Time Frame: 48 hours post-baseline (Follow-up 1)
Population: Data were not collected, as planned analysis could not be performed due to early study termination.
Groups:
- Saline: Non-Enhanced Computed Tomography (NECT): Participants received 1 intravenous injection of saline placebo (matched to Visipaque™) and underwent CT examination and supplemental non-contrast duplex ultrasonography imaging examination.
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Assessment of the Incidence of Acute Kidney Injury (AKI) Stage >=2 Per Acute Kidney Injury Network (AKIN) Serum Creatinine (SCr) Criteria
Description: as for outcome 1
Time Frame: 48 hours post-baseline (Follow-up 1)
Population: Data were not collected, as planned analysis could not be performed due to early study termination.
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Assessment of the Incidence of Acute Kidney Injury (AKI) by Contrast Induced Nephropathy (CIN)
Description: Standard definition of CIN: Increase in SCr of 0.5 mg/dL or more in the 24 to 72 hours after the CT scan.
Time Frame: 48 hours post-baseline (Follow-up 1)
Population: Data were not collected, as planned analysis could not be performed due to early study termination.
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Assessment of the Incidence of Acute Kidney Injury (AKI) Stage >=2 By Waikar Criteria
Description: Waikar's definitions of AKI: Stage 1: 0.3 mg/dL increase in SCr over 24 hours or a 0.5 mg/dL increase in SCr over 48 hours. Stage 2: 0.5 mg/dL increase in SCr over 24 hours or a 1.0 mg/dL increase in SCr over 48 hours. Stage 3: 1.0 mg/dL increase in SCr over 24 hours or a 1.5 mg/dL increase in SCr over 48 hours.
Time Frame: 48 hours post-baseline (Follow-up 1)
Population: Data were not collected, as planned analysis could not be performed due to early study termination.
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: All Cause Mortality and Morbidity
Description: Mortality (all cause death) and morbidity i.e. critical events.
Time Frame: From Baseline to Month 6
Population: Data were not collected, as planned analysis could not be performed due to early study termination.
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Blinded Independent Assessment of Image Quality/Diagnostic Confidence Using a 5-Point Scale
Description: Blinded independent assessment of image quality/diagnostic confidence using a 5-point scale. Image quality/diagnostic confidence for all imaging studies was rated on a 5-point scale from 1 (poor) to 5 (excellent).
Time Frame: Month 6
Population: Data were not collected, as planned analysis could not be performed due to early study termination.
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from randomization until the end of the follow-up period (Month 6) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are study-emergent AEs that is AEs that developed/worsened during any time after randomization until end of the follow-up period (Month 6). Analysis was performed on safety population which included all participants who were randomized to receive Visipaque™ or saline placebo and had post-randomization observations.
Arm/Group | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) | Saline: Non-Enhanced Computed Tomography (NECT)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visipaque™: Contrast-Enhanced Computed Tomography (CECT) (N=2) | Saline: Non-Enhanced Computed Tomography (NECT) (N=2)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was early terminated after enrollment of 4 participants due to very slow recruitment rates. Sample size was 4 participants instead of planned 1164 participants, hence no statistical analyses were performed, no tables and listings were produced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT03119662/Prot_SAP_000.pdf